CLINICAL TRIAL: NCT03809988
Title: International,Multicenter,Randomized,Open-label, Phase II to Evaluate the Efficacy and Safety of Continuation of Palbociclib+2nd Line Endocrine Therapy in HR+/HER2- ABC Patients Who Had Clinical Benefit During 1st Line Palbociclib.
Brief Title: PALbociclib Rechallenge in horMone Receptor-posItive/HER2- Negative Advanced Breast Cancer (PALMIRA)
Acronym: PALMIRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP068; 2017-002781-48 (EudraCT Number)
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer; Advanced Breast Cancer; Hormone Receptor Positive Tumor; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast
Keywords: HR; breast cancer; ABC; progesterone receptor; HER2; advanced; estrogen receptor
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Letrozole; Fulvestrant

STUDY DESIGN:
Intervention Model Description: Randomized 2:1
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Arm (Arm A) (Experimental): Patients will receive palbociclib capsules orally once daily (QD) (at 100mg or 125mg depending on previous treatment dose) for 21 days every four weeks in combination with endocrine therapy (letrozole or fulvestrant).
  Interventions: Drug: Palbociclib; Drug: Endocrine therapy
- Control Arm (Arm B) (Active Comparator): Patients will receive endocrine therapy (letrozole or fulvestrant).
  Interventions: Drug: Endocrine therapy

INTERVENTIONS:
Drug: Palbociclib — Palbociclib capsules orally once daily (QD) (at 100mg or 125mg depending on previous treatment dose) for 21 days every four weeks
  Other Names: IBRANCE
  Arms: Interventional Arm (Arm A)
Drug: Endocrine therapy — Endocrine therapy alone (letrozole or fulvestrant)
  Other Names: letrozole; fulvestrant

SUMMARY:
Hormone Receptor (HR)-positive/Human Epidermal Growth Factor Receptor 2 (HER2)-negative advanced breast cancer (ABC)

DETAILED DESCRIPTION:
Pre- and post-menopausal women age ≥ 18 years with HR-positive and HER2-negative with ABC that had previously received first-line endocrine therapy in combination with palbociclib and had achieved clinical benefit during palbociclib-based treatment. Patients relapsing on a palbociclib-based regimen in the adjuvant setting are also eligible. Patients are not eligible if they are candidates for a local treatment with a curative intention. Evidence of either measurable and biopsiable metastatic disease (as for Response Evaluation Criteria In Solid Tumors (RECIST v.1.1)) or non-measurable disease with bone lesion is required. Pre-menopausal women must be under treatment with luteinizing hormone-releasing hormone (LHRH) analogues.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients over 18 years of age.
2. Pre-menopausal women provided they are being treated with a LHRH analogue for at least 28 days (if shorter, post-menopausal levels of serum estradiol/Follicle-stimulating hormone (FSH) must be confirmed analytically) prior to study entry or post- menopausal women as defined by any of the following criteria:

   1. Age ≥60 years;
   2. Age <60 years and cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and serum estradiol and/or FSH level within the laboratory's reference range for postmenopausal females;
   3. Documented bilateral oophorectomy.
3. Eastern Cooperative Oncology Group (ECOG) performance status lower or equal to 1.
4. Life expectancy greater or equal to 12 weeks.
5. Histologically proven diagnosed of ABC not amenable to curative treatment.
6. Documented recurrent ER-positive and/or progesterone receptor (PgR)-positive (with ≥1% positive stained cells (according to NCCN National Comprehensive Cancer Network and ASCO American Society of Clinical Oncology guidelines) and HER2-negative (0-1+ by immunohistochemistry (IHC) or 2+ and negative by in situ hybridization (ISH) test) breast cancer in the advanced setting.
7. Radiological or clinical evidence of disease progression on first- line combination of palbociclib plus endocrine therapy (aromatase inhibitor (AI) or fulvestrant). Patients previously treated with the combination of palbociclib and tamoxifen will be excluded.
8. Patients have achieved clinical benefit criteria to a first-line palbociclib-based endocrine regimen (defined as at least stable disease ≥ 24 weeks or partial or complete response confirmed or unconfirmed).
9. Patients must have been treated with a stable minimum dose of 75 mg palbociclib during the last 2 cycles of the prior palbociclib-based regimen.
10. Last dose of palbociclib administered not later than 8 weeks and not earlier than 7 days from study entry, with the exception of patients relapsing on a palbociclib-based regimen in the adjuvant setting.
11. Patients should not have been treated in the advanced setting with at least one of these endocrine therapy options: either fulvestrant or AI.
12. Patients must have measurable disease or evaluable disease according to RECIST criteria v.1.1. Patients with only bone lesions are eligible.
13. Willingness and ability to provide tumor biopsy (if feasible) both at the time of the inclusion and after disease progression in order to perform exploratory studies. If not feasible, patient eligibility should be evaluated by a Sponsor's qualified designee.
14. Patients agree to collection of blood samples (liquid biopsy) at the time of inclusion, after 2 weeks of treatment, and upon progression or study termination.
15. Adequate organ function: (Hematological, hepatic and renal)
16. Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
17. Patients have been informed about the nature of study, and have agreed to participate in the study, and signed the informed consent form prior to participation in any study-related activities.
18. Resolution of all acute toxic effects of prior anti-cancer therapy to grade 1

Exclusion Criteria:

1. HR or HER2 unknown disease.
2. HER2-positive disease based on local laboratory results (performed by IHC / ISH test).
3. Locally ABC candidate for curative treatment.
4. Formal contraindication to endocrine therapy defined as visceral crisis and rapidly or symptomatic progressive visceral disease.
5. Prior therapy with any other CDK4/6 inhibitor different from palbociclib.
6. Known active uncontrolled or symptomatic Central Nervous System (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth. Patients with a history of CNS metastases or cord compression are eligible if they have been definitively treated and are clinically stable off anticonvulsants and steroids for at least 4 weeks before randomization.
7. Patients are currently receiving food or drugs known to be strong inducers or inhibitors of CYP3A4.
8. Current or prior malignancy which could affect compliance with the protocol or interpretation of results. Patients with curatively- treated non-melanoma skin cancer, non-muscle-invasive bladder cancer, or carcinoma in situ, among others, are generally eligible.
9. No other systemic therapy for metastatic disease including chemotherapy, immunotherapy, targeted therapy (small molecules/ monoclonal antibodies), or endocrine therapy excluding first-line palbociclib-based regimen.
10. Major surgery (defined as requiring general anesthesia) or significant traumatic injury within 2 weeks of start of study drug, or patients who have not recovered from the side effects of any major surgery, or patients who may require major surgery during the study.
11. Radiotherapy or limited-field palliative radiotherapy within 7 days prior to study enrolment, or patients who have not recovered from radiotherapy-related toxicities to baseline or grade ≤ 1 and/or from whom ≥ 25% of the bone marrow has been previously irradiated.
12. Use of concurrent investigational agents or other concomitant anticancer therapies.
13. Active bleeding diathesis, previous history of bleeding diathesis, or chronic anti-coagulation treatment (the use of low molecular weight heparin is allowed as soon as it is used as prophylaxis intention).
14. Serious concomitant systemic disorder (e.g., active infection including HIV, or cardiac disease) incompatible with the study (at the discretion of investigator).
15. Unable to swallow capsules or tablets.
16. History of malabsorption syndrome or other condition that would interfere with enteral absorption.
17. Any of the following within 6 months of randomization:

    myocardial infarction, severe/unstable angina, ongoing cardiac dysrhythmias of NCI-CTCAE v.5.0 grade ≥2, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident including transient ischemic attack, or symptomatic pulmonary embolism.
18. Uncontrolled electrolyte disorders of NCI-CTCAE v.5.0 grade ≥ 2.
19. Known hypersensitivity to palbociclib or any of its excipients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
PFS (Progression-free survival) | Baseline up to 29 months
  From a clinical point of view, the primary endpoint for this study is the PFS (progression-free survival) - defined as the period of time from randomization until objective tumor progression or death - assessed by RECIST criteria v.1.1, of continuation of palbociclib treatment combined with second-line endocrine therapy (letrozole or fulvestrant) versus endocrine therapy in pre- and post- menopausal women with HR-positive/HER2-negative ABC.

SECONDARY OUTCOMES:
Safety AEs | Baseline up to 29 months
  Patient safety and adverse events (AEs) will be evaluated using the NCI-CTCAE v.5.0. Grade 3 and 4 AEs and serious adverse events (SAEs) will be assessed to determine the safety and tolerability of the different treatment arms.
Efficacy (ORR) | Baseline up to 29 months
  To compare the objective response rate (ORR), the duration of response (DoR), the time to response (TTR), the clinical benefit rate (CBR), the time to progression (TTP), and the overall survival (OS) of palbociclib plus second-line endocrine therapy (letrozole or fulvestrant) versus endocrine therapy alone
Efficacy (Quality of Life) | Baseline up to 42 months
  To compare the patient reported global Quality of Life (QOL), functioning and symptoms of palbociclib plus second-line endocrine therapy (letrozole or fulvestrant) versus endocrine therapy alone.
Efficacy of subgroup analysis | Baseline up to 42 months
  To perform subgroup analysis for primary and secondary endpoints in stratified groups of patients.
Compare efficacy | Baseline up to 42 months
  To compare the time to first chemotherapy of palbociclib plus second-line endocrine therapy (letrozole or fulvestrant) versus endocrine therapy alone.
Exploratory objectives (molecular markers) | Baseline up to 42 months
  To explore potential molecular markers of sensitivity and/or resistance for the combination and endocrine therapy alone, according to, but not limited to, the results obtained from the BioPER trial (NCT03184090).
Exploratory objectives (intrinsic molecular subtypes) | Baseline up to 42 months
  To explore correlations between the intrinsic molecular subtypes and efficacy/safety findings in patients with HR-positive/HER2- negative ABC.

CONTACTS AND LOCATIONS:
Overall Officials: José Perez, Principal Investigator — MedSIR
Locations (53):
- France (7):
  - Hôpital Jean Minjoz, Besançon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - CHD Vendee, La Roche-sur-Yon
  - Hopital Europeen Georges Pompidou, Paris
  - Hôpital Tenon AP-HP, Paris
  - Centre Paul Strauss, Strasbourg
- Germany (8):
  - University Hospital Dresden-GYN, Dresden
  - Kliniken Essen Mitte, Essen
  - Universitätsklinikum Essen Frauenklinik, Essen
  - AGAPLESION Markus Krankenhaus, Frankfurt
  - Technical University Munich, Munich
  - UKM Brustzentrum, Münster
  - Klinikum Ernst von Bergmann, Potsdam
  - Klinikum Mutterhaus der Borromäerinnen Trier, Trier
- Italy (4):
  - Ospedale Civili Brescia, Brescia
  - Instituto Europeo di Oncologia, Milan
  - Oncologia Medica Ospedale di Prato, Prato
  - Policlinico Universitario Campus Bio-medico, Roma
- Slovenia (2):
  - Onkološki Inštitut Ljubljana, Ljubljana
  - Univerzitetni klinicni center Maribor Oddelek za onkologijo, Maribor
- Spain (26):
  - ICO Badalona, Badalona, Barcelona
  - Hospital Provincial de Castellón, Castelló, Castelló
  - Consorci Sanitari de Terrassa, Terrassa, Terrasa
  - Centro Oncológico de Galicia, A Coruña
  - Institut Català d'Oncologia Bellvitge, Barcelona
  - H. Vall Hebrón, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital San Pedro de Alcantara, Cáceres
  - Institut Català d'Oncologia, Girona
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Sanchinarro, Madrid
  - Hospital La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Sant Joan, Reus
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Instituto Valenciano de Oncología IVO, Valencia
  - Hospital General Universitari de Valencia, Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Álvaro Cunqueiro, Vigo
  - Hospital Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza
- United Kingdom (6):
  - Darent Valley Hospital by Dartford and Gravesham NHS Trust, Dartford
  - Beatson West of Scotland Cancer Center, Glasgow
  - Barts Cancer Institute, London
  - Kent Oncology Department, Maidstone
  - Abertawe Bro Morgannwg University Local Health Board, Singleton Hospital, Swansea
  - Royal Cornwall Hospital NHS Trust, Truro

IPD SHARING:
Plan to Share IPD: Yes
Study Leaflet V2_20190115 with study design, primary objetive, inclusion criteria and exclusion criteria
Supporting Information: Study Protocol
Time Frame: During recruitment period
Access Criteria: Oncology department

REFERENCES:
- [Derived] Llombart-Cussac A, Harper-Wynne C, Perello A, Hennequin A, Fernandez-Ortega A, Colleoni M, Marin S, Quiroga V, Medioni J, Iranzo V, Wheatley D, Del Barco Berron S, Anton A, Dobi E, Ruiz-Borrego M, Alcala-Lopez D, Perez-Escuredo J, Antonarelli G, Sampayo-Cordero M, Perez-Garcia JM, Cortes J. Second-Line Endocrine Therapy With or Without Palbociclib Rechallenge in Patients With Hormone Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: PALMIRA Trial. J Clin Oncol. 2025 Jun 20;43(18):2084-2093. doi: 10.1200/JCO-24-01865. Epub 2025 Apr 28. PMID 40294349